CLINICAL TRIAL: NCT04671849
Title: An Open Label, Multi-center, Phase I Clinical Study to Evaluate the Safety, Effectiveness and Pharmacokinetic Characteristics of SIM1803-1A in Patients With Locally Advanced/Metastatic Solid Tumors With NTRK, ROS1 or ALK Gene Fusion Mutations.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM1803-1A-NTRK-0101
Record Dates: First submitted 2020-12-15; First posted 2020-12-17 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Advanced or Metastatic Solid Tumors With NTRK, ROS1 or ALK Gene Fusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- adult patients_Dose 1 (Experimental)
  Interventions: Drug: SIM1803-1A
- adult patients_Dose 2 (Experimental)
  Interventions: Drug: SIM1803-1A
- adult patients_Dose 3 (Experimental)
  Interventions: Drug: SIM1803-1A
- adult patients_Dose 4 (Experimental)
  Interventions: Drug: SIM1803-1A
- adult patients_Dose 5 (Experimental)
  Interventions: Drug: SIM1803-1A
- adult patients_Dose 6 (Experimental)
  Interventions: Drug: SIM1803-1A
- adult patients_Dose 7 (Experimental)
  Interventions: Drug: SIM1803-1A
- adult patients_Dose 8 (Experimental)
  Interventions: Drug: SIM1803-1A

INTERVENTIONS:
Drug: SIM1803-1A — SIM1803-1A will be administered orally as tablets at a given dose once daily in continuing 21-days cycles.

SUMMARY:
This research study is done to test the safety, effectiveness and pharmacokinetic characteristics of SIM1803-1A in patients with locally advanced/metastatic solid tumors with NTRK, ROS1 or ALK gene fusion mutations. The cancer must have a change in a particular gene (NTRK1, NTRK2, NTRK3, ROS1 or ALK). SIM1803-1A is a drug that blocks the actions of these NTRK/ ROS1 /ALK genes in cancer cells and can therefore be used to treat cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a locally advanced or metastatic solid tumor that has progressed or was nonresponsive to available therapies, are unfit for standard chemotherapy or for which no standard or available curative therapy exists；Proof of a malignancy harboring a NTRK、ROS1 or ALK fusion；Eastern Cooperative Oncology Group (ECOG) score of 0 or 1 and a life expectancy of at least 3 month；Adequate hematologic, hepatic, and renal function；Signed informed consent form；

Exclusion Criteria:

* Any contraindications as listed in the local approved product information；Patients with unstable primary central-nervous-system tumors or metastasis, exceptions possible；Pregnancy or lactation；Clinically significant active cardiovascular disease or history of myocardial infarction；Participation in an investigational program with interventions outside of routine clinical practice；Prior treatment with other kinase inhibitor with tropomyosin receptor kinase inhibition；Active uncontrolled systemic bacterial, viral, or fungal infection；Current treatment with a strong CYP3A4 inhibitor or inducer；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 5 years
  Number of participants with adverse events
Severity of adverse events | 5 years
  Severity of adverse events
Maximum tolerated dose | 5 years
  Maximum tolerated dose
Recommended dose for dose expansion | 5 years
  Recommended dose for dose expansion
Maximum concentration of SIM1803-1A in plasma (Cmax) | Predose and 0.25, 0.5, 1, 2, 4, 8，12，24and 48 hours after drug administration on Days 1 and 8 of Cycle 1（each cycle is 21 days）
  Maximum concentration of SIM1803-1A in plasma (Cmax)
Area under the concentration-time curve of SIM1803-1A in plasma from time 0 to 24 hours in fasted state (AUC(0-24)_fasted) | Up to 1 day
  Area under the concentration-time curve of SIM1803-1A in plasma from time 0 to 24 hours in fasted state (AUC(0-24)_fasted)
Area under the concentration-time curve of SIM1803-1A in plasma from time 0 to infinity in fasted state (AUC_fasted) | Up to 3 days
  Area under the concentration-time curve of SIM1803-1A in plasma from time 0 to infinity in fasted state (AUC_fasted)
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 24 weeks
  Number of participants with treatment-emergent adverse events (TEAEs)
Time to maximum concentration of SIM1803-1A in plasma (Tmax) | Predose and 0.25, 0.5, 1, 2, 4, 8，12，24and 48 hours after drug administration on Days 1 and 8 of Cycle 1（each cycle is 21 days)
  Time to maximum concentration of SIM1803-1A in plasma (Tmax)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 60 months
  Overall Response Rate (ORR)
Duration of Response (DOR) | Up to 60 months
  Duration of Response (DOR)
progression-free survival（PFS） | Up to 60 months
  progression-free survival（PFS）

CONTACTS AND LOCATIONS:
Overall Officials: shun lu, Ph.D, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No